CLINICAL TRIAL: NCT03063229
Title: Energy Balance Following Islet Transplantation
Acronym: EBFIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants due to lack of patients eligible at the time
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC 16/SS0031 R&D: 2016/0118
Record Dates: First submitted 2016-11-23; First posted 2017-02-24 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Pump Therapy; Islet Cell Transplant; Energy Expenditure
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Hematologic Tests; Magnetic Resonance Spectroscopy; Diet Records; Continuous Glucose Monitoring; Surveys and Questionnaires; Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Islet Transplant Patients (Active Comparator): Patients with Type 1 Diabetes who are on the waiting list to undergo an islet transplant.
  Interventions: Device: Accelerometer; Other: Anthropomentry; Procedure: Blood tests; Device: BODPOD; Procedure: MRI (Magnetic Resonance Imaging); Other: Food Diary; Device: CGMS (Continuous Glucose Monitoring System); Other: Questionnaire and Hypo Score; Procedure: Mixed Meal Tolerance Test (MMTT); Procedure: Indirect Calorimetry; Drug: Doubly Labelled Water; Drug: Hepatic Mitochondrial Oxidation breath test
- Insulin Pump Therapy Patients (Active Comparator): Patients with Type 1 Diabetes waiting to start on an Insulin Pump.
  Interventions: Device: Accelerometer; Other: Anthropomentry; Procedure: Blood tests; Device: BODPOD; Procedure: MRI (Magnetic Resonance Imaging); Other: Food Diary; Device: CGMS (Continuous Glucose Monitoring System); Other: Questionnaire and Hypo Score; Procedure: Mixed Meal Tolerance Test (MMTT); Procedure: Indirect Calorimetry; Drug: Doubly Labelled Water; Drug: Hepatic Mitochondrial Oxidation breath test
- Healthy Volunteers (Other): Participants with no Diabetes.
  Interventions: Device: Accelerometer; Other: Anthropomentry; Procedure: Blood tests; Device: BODPOD; Other: Food Diary; Device: CGMS (Continuous Glucose Monitoring System); Procedure: Mixed Meal Tolerance Test (MMTT); Procedure: Indirect Calorimetry

INTERVENTIONS:
Device: Accelerometer — Attach a monitor to participants thigh to measure their physical activity for 7 days. The monitor is called the Activpal Micro.
  Other Names: Activpal Micro
Other: Anthropomentry — Take skinfold measurements of participants using Harpenden skinfold calipers.
Procedure: Blood tests — Taking standard clinical blood tests to measure HbA1c, Glucose, FBC, U&E's, LFT's, Coagulation Screen, Lipid Profile, Thyroid Function, and Tacrolimus for transplant patients.
Device: BODPOD — Measure body composition using a BODPOD machine. This uses Air displacement plethysmography.
Procedure: MRI (Magnetic Resonance Imaging) — MRI Scans of abdomen, particularly the livers of islet transplant and insulin pump patients.
  Arms: Insulin Pump Therapy Patients; Islet Transplant Patients
Other: Food Diary — Participants will keep a 7 day weighed food diary.
Device: CGMS (Continuous Glucose Monitoring System) — Participants will wear a CGMS for 7 days to measure their glucose control and pattern over a 7 day period.
Other: Questionnaire and Hypo Score — Participants with Type 1 Diabetes will fill in 3 short questionnaires about their Diabetes.
  Other Names: Clark and Gold Score and Fear of Hypo Survey
  Arms: Insulin Pump Therapy Patients; Islet Transplant Patients
Procedure: Mixed Meal Tolerance Test (MMTT) — The patients will under go a test which involves taking 30 minute glucose and C-peptide levels (blood test from a cannula) for 3 hours. They will consume 150ml of a mixed meal supplement drink "Fortisip Compact" at the start of the 3 hours, after having no morning insulin, breakfast and not eating anything from midnight the night before.
Procedure: Indirect Calorimetry — During the Meal Tolerance Test, the patients will be resting on a bed in the research facility and breathing normally into a clear plastic hood. The machine connected to the hood (GEM) will analyse their resting energy expenditure from the gases expired in their breath. They will have the hood on for 2 hours.
  Other Names: GEM
Drug: Doubly Labelled Water — The Doubly Labelled water will be prescribed for the participants and they will drink their 100ml dose of the stable isotope. Dose depends on the eight of the participant. The participant will then collect urine samples at home on day 5, 10 and 14 after drinking the water. They will store them in the freezer until they can bring them back to us.
  Arms: Insulin Pump Therapy Patients; Islet Transplant Patients
Drug: Hepatic Mitochondrial Oxidation breath test — Participants will be given a calculated amount of the stable isotope C-Octanoate, which will be delivered in a water solution. They will then be asked to breath down a small tube into a clear plastic collection bag 10 times over 2 hours.
  Other Names: IRIS machine.
  Arms: Insulin Pump Therapy Patients; Islet Transplant Patients

SUMMARY:
Islet transplantation may be appropriate in up to 10% of adults with Type 1 diabetes who suffer repeated episodes of hypoglycaemia with severely impaired awareness of hypoglycaemia (IAH) (1). Our Scotland-wide islet transplant programme performed its first transplant in February 2011 and 30 islet transplants have followed in 18 recipients. Following islet transplantation we have observed improved glycaemic control in all subjects. When metabolic control is improved with exogenous insulin, weight gain is common (2). In our transplant recipients significant reductions in bodyweight and fat mass with no significant reduction in total caloric intake pre- versus post-transplantation has been observed. We hypothesise that energy expenditure is increased post-transplantation leading to weight loss and diminished fat mass. The mechanisms that may be implicated include increased activity energy expenditure, increased resting energy expenditure (REE) and, or, increased post-prandial thermogenesis (PPT= the energy expended after a meal) secondary to increased portal circulation of insulin being partially or fully restored, and diminished circulating systemic insulin concentrations with a decreased propensity for storing fat. The aim of this study is to understand the mechanism of weight loss and body compositional changes by detailed examination of energy intake and energy expenditure in transplant recipients along with control subjects listed for insulin-pump therapy and glucose tolerant controls. These detailed studies are lacking in islet transplantation and are important as they will reveal how physiology is altered post-transplantation, if peripheral hyperinsulinaemia (insulin-pump subjects and pre-transplant subjects) negatively affects energy expenditure and how quantitative measures such as activity energy expenditure, diet and quality-of-life measures such as fear of hypoglycaemia alter post-transplant. This will lead to the improved management of patients with hypoglycaemia and IAH.

DETAILED DESCRIPTION:
Background and rationale for the study: Type 1 Diabetes, Hypoglycaemia, IAH and Islet Transplantation

Type 1 diabetes is caused by autoimmune destruction of beta cells within the islets of the pancreas. Those with Type 1 diabetes are dependent on daily insulin replacement for survival and despite major advances in treatment (3), life-expectancy is reduced significantly due to metabolic crises and increased risk of major atherosclerotic vascular events (4). All complications of chronic high glucose can be prevented by tight glycaemic control (5) but this is, however, counter-balanced by a high risk of severe hypoglycaemia leading to a reduced ability to perceive the onset of hypoglycaemia, with disabling confusion and collapse without warning, termed Impaired A Awareness of Hypoglycaemia (AIH). IAH affects up to 25% of people with established Type 1 diabetes every year (10-15 million people world-wide) (6, 7). Approximately 30,000 people in Scotland have Type 1 diabetes and the prevalence is increasing (8). Those with recurrent hypoglycaemia with severe IAH, often experience fluctuations in blood glucose and may be eligible for islet transplantation (5). Islets are transplanted in high numbers via the portal vein under radiological guidance into the liver with glucocorticoid free immunosuppression ("Edmonton protocol"). Two or more transplants are usually necessary to regain insulin secretion to allow adequate control of glucose concentrations and restore awareness of hypoglycaemia.

UK Islet Transplant Consortium (UKITC), Scottish National Islet Programme and anthropometric changes post islet transplantation

Our transplant programme is one of seven in the UKITC; other sites include Newcastle, Oxford, London (Kings, Royal Free), Manchester and Bristol. The primary goal in the UK is to reduce the frequency and restore awareness of hypoglycaemia. Referred patients are assessed in depth by a multidisciplinary team pre-transplant, at the time of transplant and then serially post-transplant. In the UK from April 2008-September 2013 there have been 96 transplants in 76 recipients. Graft survival is >88%, as defined by a stimulated c-peptide of >100pmol/L (90 min following a Fortisip meal), and there have been significant decreases in the frequency of hypoglycaemia: pre- vs. post-transplant, median (interquartile range): 21(7-79) vs. 0(0-1) episodes of hypoglycaemia per annum with significant reductions in HbA1c and insulin dose (all p<0.01)(9). Body weight at 1 year in the UKITC cohort is significantly diminished; pre-transplant: mean (±SEM) 66.3(±1.2) vs. 62.3(±1.1) kg (p=0.001). In common with many programmes (10) peak function is seen at 3 months following the first transplant often with insulin independence but a variable degree of attrition in function may be seen following this with many patients on insulin 1 year following their transplant, although at a much reduced dose versus pre-transplant. In Scotland we have performed 47 transplants in 29 recipients. Those patients with Type 1 diabetes and normal renal function have been assessed previously (≥3<30 months) post-transplant (n=14; 6 males, 8 females; age (range: 30-57 years); all have functioning grafts. Following islet transplantation we have observed significant reductions in body weight, pre versus post-transplant: median(interquartile range) 70.9(64.9-82.5) vs. 66.0(59.8-79.9)kg, p=0.01; BMI: 26.2(24.4-28.6) vs. 24.5(22.2-26.1) kg/m2, p=0.01; %fat mass: 30.0(21.2-35.2) vs. 24.1(18.4-31.2)%, p=0.004; and waist circumference: 85.5(77-89.7) vs. 77.5(73.5-88.3)cm, p=0.01. Total calorific intake assessed via 7 day dietary histories were not different pre- versus post-transplant 1700(1581-1842) vs. 1528(1319-1708) kcal, (p=0.09), although frequency of hypoglycaemia (10(6-18) vs 1(0-3)) episodes per week and calorific intake for hypoglycaemia were reduced. Concurrently HbA1c has improved p<0.001 (11).

Consistent with our observations, significant reductions in body weight of >4kg (10, 12), waist circumference and body fat mass, the latter measured using bioelectrical impedence, within a year of islet transplantation, have been previously reported, despite no significant changes in caloric intake post-transplant (12). In the latter study 30 subjects had all assessments completed and 12 subjects were not on insulin at the time of their last data collection. Insulin use reduced 10 fold and glycaemic control improved. Regression analyses adjusting for confounding variables including exogenous insulin dose and glucagon-like peptide-1 agonist use, confirmed the association of weight loss with islet transplantation. Of note in this cohort of islet transplant recipients, no measurements of energy expenditure were made and the patients including those with islet transplants following kidney transplants were on a variety of immunosuppressant agents which may affect energy balance. More recently the same group published a retrospective study in islet transplant recipients and found a decrease in BMI in their cohort of 33 recipients at 3 years post-transplant versus pre-transplant (13). Dietetic habits and caloric intake and activity, both assessed by open ended questionnaires, were not significantly altered pre- versus post-transplant.

We hypothesise that other components of energy expenditure are increased following islet transplantation secondary to the diminished ratio of systemic to portal insulin concentrations. The energy expenditure components that may be modulated in this way include REE and PPT.

Our proposed study aims to prospectively assess energy intake and food choices using the "gold standard" of serial 7 day weighed food diaries (14, 15) and assess the multiple components of energy expenditure pre- and post-islet transplantation versus subjects commencing insulin pump therapy who have relatively high ratios of systemic to portal insulin concentrations along with control subjects with normal glucose tolerance.

Maintenance of body weight and relationship with energy intake and energy expenditure

Bodyweight reflects the balance between food intake and energy expenditure. Total energy expenditure may be separated into three main components: REE, PPT and physical activity. REE may be defined as energy expenditure at rest in the fasted state measured in a thermoneutral environment. PPT or diet induced thermogenesis is an increase in metabolic rate above REE; PPT demonstrates more variability between people than REE (16, 17). It is the energy generated following food ingestion and has an obligatory component reflecting the energy required to digest, absorb, interconvert and store fuels and a facultative component in which the sympathetic nervous system has a major role (17). The increment in energy expenditure may be accounted for in part by the cost of glucose storage as glycogen but often the measured cost of glucose storage is much higher than this and it is this increment above this "obligatory component" that is termed "facultative thermogenesis" (18). This facultative component can compromise 50% of the thermic effect of food and large inter individual variations may be present (19, 20). With a sedentary lifestyle, REE constitutes 75 to 80%, PPT 10 to 15% and physical activity 10 to 15% of total daily energy expenditure.

Modulators of energy expenditure

The lean body mass, thyroid status and protein turnover of a subject determines the REE (21). We and others have shown that PPT is negatively related to insulin sensitivity in a group at risk for Type 2 diabetes (22). PPT may be affected by beta-adrenergic blockade and other drugs (23, 24). Insulin, a known vasodilator, may also affect energy expenditure (25). Intraportally transplanted islets may become revascularised by tributaries from both the portal vein and the hepatic artery (26) or perhaps by tributaries from just the hepatic artery (27). It is untested if PPT increases as a consequence of islet transplantation secondary to increased insulin concentrations in the portal and splanchnic circulations (28). There has been much progress in the induction agents and immunosuppression therapy used over the last 10 years with improved insulin independence rates (29). Our centre uses the monoclonal antibody alemtuzumab at induction (30) and maintenance immunosuppression is with the calcineurin inhibitor tacrolimus and mycophenolate. Liver transplant patients on tacrolimus have diminished REE, suggesting an inhibition of mitochondrial respiration (31) although in liver transplantation hepatic denervation occurs with autonomic nerve dysfunction which may also decrease energy expenditure (32, 33). It is unlikely therefore that the immunosuppressive therapies increase energy expenditure although there may certainly be negative effects on appetite and energy intake (34).

Hepatic fatty acid oxidation.

Free Fatty Acids (FFA) are oxidised within mitochondria which are present within the whole body with large concentrations in the liver, muscle and heart. Most methodologies measure whole body fatty acid oxidation rates and cannot distinguish between these sources. Hepatic fat oxidation may be altered following islet transplantation and may influence hepatic insulin sensitivity. It is not known whether hepatic fat oxidation is increased following islet transplantation which may explain the weight loss.

Assessment of mitochondrial fatty acid oxidation in the liver:

The assessment of hepatic mitochondrial function has been hampered by invasive and complex techniques, which have in general lacked specificity. Recently, breath testing using stable carbon isotopes has been proposed as a safe, non-invasive and non-radioactive method to assess mitochondrial oxidative capacity. Sodium13C-octanoate can be employed as a substrate used in assessing hepatic mitochondrial oxidative function, particularly, β-oxidative pathway. Sodium octanoate is a medium chain fatty acid, which is metabolised through mitochondrial β-oxidation, producing acetyl Coenzyme A (acetyl Co-A). Acetyl Co-A enters the Krebs cycle to undergo further oxidation leading to the production of CO2 that can be measured during the breath test (35a).

The purpose of this proposal is to understand the mechanisms of the weight loss and fat mass observed. No study has examined energy expenditure prospectively in this detailed way in a cohort of pre- and post-islet transplant and insulin pump therapy recipients.

Detailed plan of investigation:

Hypothesis: Islet transplantation is associated with increased energy expenditure as a consequence of the reduction in the ratio of systemic to portal insulin concentrations.

The aims are to assess:

1. Anthropometric measures: body weight, waist circumference, skin fold thickness, body composition using air displacement plethysmography (Bod Pod).
2. Total energy intake, including the excess energy intake required in the treatment of hypoglycaemia, using 7 day weighed food diaries, The Fear of Hypoglycaemia Survey, Gold and Clarke Score.
3. The activity component of energy expenditure using accelerometry.
4. REE and PPT (using meal tolerance tests) and total metabolic rate (TMR) using doubly labelled water.
5. Hepatic fat oxidation using Sodium 13C octanoate.
6. Liver fat, abdominal subcutaneous and visceral fat using MRS and MRI.

In the islet transplant recipients and insulin pump patients MRS of liver and MRI of liver fat; abdominal subcutaneous and visceral fat; glycaemic lability; frequency of hypoglycaemia assessed using continuous glucose monitoring systems (CGMS); awareness of hypoglycaemia assessed subjectively with the Gold Score and Clarke Scores (35), and mixed meal tolerance tests will continue as per the UKITC protocols, including pre-transplantation. In the glucose tolerant controls all the above will be done except the MR imaging studies, the Fear of Hypoglycaemia Survey (36), the Gold and Clarke scores and CGMS.

STUDY DESIGN In the islet transplant programme recipients are assessed pre-transplant and at 1, 3, 6, 12 months post-transplant and then 6 monthly. The investigations in the transplant or insulin pump subjects, will be based around these timelines. Specifically, we anticipate peak islet function at 3 months.

We aim to recruit 3 groups of participants: those with Type I diabetes that are on the waiting list for islet transplantation, those with Type I diabetes that are on the waiting list for insulin pump therapy, and controls who do not have diabetes (glucose tolerant).

The study contains 3 parts as described below. The participants will be expected to complete all 3 parts at each time point. The 3 parts are completed over 5 separate time points totalling 13 visits:

The following visits are for the patients with type 1 diabetes:

Pre- intervention and then 1,3, 6 and 12 months post intervention.

* Pre-intervention there are 3 study visits over a 4 week period
* Month 1 post intervention there are 2 visits over 2 weeks
* Months 3 post invention there are 3 visits over a 4 week period
* Month 6 post intervention there are 2 visits over 2 weeks
* 12 months post intervention there are 3 visits over 4 weeks

Patients with diabetes normally have 1 routine clinic visit at each time point described as part of their normal follow-up post-intervention. The other visits will be surplus to their usual follow-up following intervention, apart from during their first month post-intervention where they would be followed-up weekly.

Glucose-tolerant controls will only have one set of examinations carried out which will involve 3 visits over 4 weeks.

Pre-intervention, 3 & 12 months

Part 1:

Blood tests (FBC, LFTS, U&Es, Coagulation Screen, Lipid Profile, Thyroid function,HbA1c, Glucose, post-transplant Tacrolimus level) this is approx 18ml (3 ½ teaspoons). This is part of the routine follow-up for islet transplant patients.

Anthropometry -body weight, waist, calf and arm circumference, skin fold thickness (including bicep, tricep, scapula, illiac crest and calf), body composition using air displacement plethysmography (BODPOD). These examinations are study specific and not part of the routine follow-up.

A continuous glucose monitoring (CGMS) device and accelerometer will also be fitted to measure energy expenditure over seven days. The participant will be given a food diary and a set of weighing scales to record food intake over this seven day period (including the excess calories required in the treatment of hypoglycaemia) at home. CGMS is frequently used during the follow-up of patients with diabetes. Glucose tolerant controls will not have a CGMS fitted or complete the following surveys.

The participant will complete "The Fear of Hypoglycaemia Survey". This is a questionnaire asking how/whether they modify their behaviour in order to avoid hypoglycaemia and how frequently they worry about their hypoglycaemia in different circumstances. The participants will also be asked about their degree of impaired awareness of hypoglycaemia using specific scoring systems (Gold and Clarke Score).

Subjects within the islet transplant cohort and pump therapy cohort will be asked to go to the clinical research imaging centre and will have magnetic resonance scanning done of their abdomen including their liver and their abdominal fat.

Part 2 (week 2):

The participant will be invited back a week later to assess their resting energy expenditure (REE). At this visit all the equipment from week 1 will be returned. The participant will be weighed on arrival and have a cannula inserted into an arm. Blood samples for glucose, insulin and c-peptide will be taken (15mls). The participants will then be given a "mixed meal" in the form of "Fortisip concentrate" which tastes like a milk shake. Their energy expenditure after this mixed meal will be measured for two hours by a device called an indirect calorimeter which is an open hood ventilation device which measures the amount of oxygen breathed in and the amount of carbon dioxide breathed out. The energy expended after a meal is called post-prandial thermogenesis (PPT) and represents the calories burnt after a meal. Simultaneously blood samples will be taken every 30 minutes for three hours to measure insulin, c-peptide and glucose levels (150 mls). This is the gold standard test for assessing islet function.

"Doubly-labelled Water" studies will be carried out on a proportion of participants. The participant will be given "doubly labelled water" to drink at their second visit, a urine sample will be collected just prior to drinking the water and then they will be instructed to collect further urine samples at home on day 1, 5, 10 and 14 following this, the research nurse will call them regularly during this time period. The samples will be stored in the freezer in a zip locked bag contained in a plastic tub with tight-fitting lid.

Part 3 (week 4):

The participant will be invited back two weeks after part 2 for a study specific visit. The urine samples will be collected. Hepatic Mitochondrial studies will carried out this involves the participant drinking a solution containing Sodium 13C Octanoate which is a fatty acid found in foods. They will then be asked to blow into a bag intermittently over a period of two hours (0, 10, 15, 20, 25, 30, 40, 60, 90 and 120 mins) in order to measure how their liver handles the fatty acid and whether they "burn" it quickly or slowly.

1 month and 6 months post intervention

Only blood test, anthropometry, accelerometer, weighed food diary and CGMS will be carried out. Islet transplant recipients will have a clinical mixed meal tolerance test carried out to assess islet function. These visits will coincide with routine visits.

ELIGIBILITY:
Inclusion Criteria:

* Islet transplant and pump therapy

  * Male or Female
  * Age 18 or over
  * Type 1 diabetes.
  * On waiting list for islet transplantation or insulin pump therapy.
  * Normal renal function (GFR >60).
  * Normal thyroid function (those on thyroxine may be included provided their thyroid function tests are normal).
  * Able to understand and undertake the study procedures.
  * Able to give signed informed consent.
* Healthy controls

  * Male or Female.
  * Age 18 or over.
  * Glucose tolerant.
  * Normal renal function (GFR >60).
  * Normal thyroid function (those on thyroxine may be included provided their thyroid function tests are normal).
  * Willingness to understand and undertake study procedures.
  * Able to give signed informed consent.

Exclusion Criteria:

* Islet transplant and pump therapy

  * Age less than 18
  * Impaired renal function (GFR <60)
  * Impaired thyroid function despite therapy
  * Unable to adhere to the study timetable.
  * Unwilling to give informed consent.
* Healthy Controls

  * Age less than 18
  * Impaired glucose-tolerance
  * Impaired thyroid function
  * Impaired renal function (GFR <60)
  * Unable to adhere to the study timetable.
  * Unwilling to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06; Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Body composition | 12 Months
  Using ISAK anthropometry methods. This includes skinfold thicknesses and waist, calf and arm circumference.
Total energy intake | 12 Months
  including the excess energy intake required in the treatment of hypoglycaemia, using 7 day weighed food diaries,
The activity component of energy expenditure using accelerometry. | 12 Months
Resting Energy Expenditure (REE) | 12 Months
  Using Indirect Calorimetry
Hepatic fat oxidation using Sodium 13C octanoate. | 12 Months
Liver fat, abdominal subcutaneous and visceral fat using MRI scans. | 12 Months
BODPOD | 12 Months
  To measure body composition using air displacement plethysmography (Bod Pod).
Hypoglycaemia scores. | 12 Months
  Fear of Hypoglycaemia Survey, Gold and Clarke Scores.
Post-Prandial Thermogenesis (PPT) | 12 Months
  Using mixed meal tolerance tests
Total metabolic Rate (TMR) | 12 Months
  Using Doubly Labelled Water

CONTACTS AND LOCATIONS:
Overall Officials: Shareen Forbes, MD, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cryer PE. Mechanisms of hypoglycemia-associated autonomic failure in diabetes. N Engl J Med. 2013 Jul 25;369(4):362-72. doi: 10.1056/NEJMra1215228. No abstract available. PMID 23883381
- [Background] Larger E. Weight gain and insulin treatment. Diabetes Metab. 2005 Sep;31(4 Pt 2):4S51-4S56. doi: 10.1016/s1262-3636(05)88268-0. PMID 16389899
- [Background] Miller RG, Secrest AM, Sharma RK, Songer TJ, Orchard TJ. Improvements in the life expectancy of type 1 diabetes: the Pittsburgh Epidemiology of Diabetes Complications study cohort. Diabetes. 2012 Nov;61(11):2987-92. doi: 10.2337/db11-1625. Epub 2012 Jul 30. PMID 22851572
- [Background] Dorman JS, Laporte RE, Kuller LH, Cruickshanks KJ, Orchard TJ, Wagener DK, Becker DJ, Cavender DE, Drash AL. The Pittsburgh insulin-dependent diabetes mellitus (IDDM) morbidity and mortality study. Mortality results. Diabetes. 1984 Mar;33(3):271-6. doi: 10.2337/diab.33.3.271. PMID 6698317
- [Background] Secrest AM, Becker DJ, Kelsey SF, LaPorte RE, Orchard TJ. All-cause mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes: the Allegheny County type 1 diabetes registry. Diabetes Care. 2010 Dec;33(12):2573-9. doi: 10.2337/dc10-1170. PMID 21115767
- [Background] Frier BM. Cognitive functioning in type 1 diabetes: the Diabetes Control and Complications Trial (DCCT) revisited. Diabetologia. 2011 Feb;54(2):233-6. doi: 10.1007/s00125-010-1983-6. Epub 2010 Nov 26. PMID 21109995
- [Background] Wright RJ, Newby DE, Stirling D, Ludlam CA, Macdonald IA, Frier BM. Effects of acute insulin-induced hypoglycemia on indices of inflammation: putative mechanism for aggravating vascular disease in diabetes. Diabetes Care. 2010 Jul;33(7):1591-7. doi: 10.2337/dc10-0013. PMID 20587725
- [Background] Govan L, Wu O, Briggs A, Colhoun HM, McKnight JA, Morris AD, Pearson DW, Petrie JR, Sattar N, Wild SH, Lindsay RS; Scottish Diabetes Research Network Epidemiology Group. Inpatient costs for people with type 1 and type 2 diabetes in Scotland: a study from the Scottish Diabetes Research Network Epidemiology Group. Diabetologia. 2011 Aug;54(8):2000-8. doi: 10.1007/s00125-011-2176-7. Epub 2011 May 24. PMID 21607632
- [Background] Brooks AM, Walker N, Aldibbiat A, Hughes S, Jones G, de Havilland J, Choudhary P, Huang GC, Parrott N, McGowan NW, Casey J, Mumford L, Barker P, Burling K, Hovorka R, Walker M, Smith RM, Forbes S, Rutter MK, Amiel S, Rosenthal MJ, Johnson P, Shaw JA. Attainment of metabolic goals in the integrated UK islet transplant program with locally isolated and transported preparations. Am J Transplant. 2013 Dec;13(12):3236-43. doi: 10.1111/ajt.12469. Epub 2013 Oct 1. PMID 24119216
- [Background] Ryan EA, Lakey JR, Paty BW, Imes S, Korbutt GS, Kneteman NM, Bigam D, Rajotte RV, Shapiro AM. Successful islet transplantation: continued insulin reserve provides long-term glycemic control. Diabetes. 2002 Jul;51(7):2148-57. doi: 10.2337/diabetes.51.7.2148. PMID 12086945
- [Background] Forbes S, McGilvray T, Davidson J, Duncan K, Jansen C, Anderson D, et al. Outcomes in subjects with Type 1 diabetes following islet transplantation in the Scottish islet transplant programme. . British Transplant Association 2012 and Diabetes UK 2013. 2013.
- [Background] Poggioli R, Enfield G, Messinger S, Faradji RN, Tharavanij T, Pisani L, Cure P, Ponte G, Baidal DA, Froud T, Ricordi C, Alejandro R. Nutritional status and behavior in subjects with type 1 diabetes, before and after islet transplantation. Transplantation. 2008 Feb 27;85(4):501-6. doi: 10.1097/TP.0b013e3181629d7b. PMID 18347527
- [Background] Delmonte V, Peixoto EM, Poggioli R, Enfield G, Luzi L, Ricordi C, Alejandro R. Ten years' evaluation of diet, anthropometry, and physical exercise adherence after islet allotransplantation. Transplant Proc. 2013 Jun;45(5):2025-8. doi: 10.1016/j.transproceed.2013.01.031. PMID 23769100
- [Background] Pears SL, Jackson MC, Bertenshaw EJ, Horne PJ, Lowe CF, Erjavec M. Validation of food diaries as measures of dietary behaviour change. Appetite. 2012 Jun;58(3):1164-8. doi: 10.1016/j.appet.2012.02.017. Epub 2012 Feb 28. PMID 22387936
- [Background] Wrieden WP, H; Armstrong, J and Barton, K. A short review of dietary assessment methods used in National and Scottish Research Studies. Working Group on Monitoring Scottish Dietary Targets Workshop. 2003.
- [Background] Jensen MD, Johnson CM, Cryer PE, Murray MJ. Thermogenesis after a mixed meal: role of leg and splanchnic tissues in men and women. Am J Physiol. 1995 Mar;268(3 Pt 1):E433-8. doi: 10.1152/ajpendo.1995.268.3.E433. PMID 7900790
- [Background] Ravussin E, Lillioja S, Anderson TE, Christin L, Bogardus C. Determinants of 24-hour energy expenditure in man. Methods and results using a respiratory chamber. J Clin Invest. 1986 Dec;78(6):1568-78. doi: 10.1172/JCI112749. PMID 3782471
- [Background] Jequier E. Carbohydrate-induced thermogenesis in man. Int J Vitam Nutr Res. 1986;56(2):193-6. PMID 3525443
- [Background] Robinson S, Niththyananthan R, Anyaoku V, Elkeles RS, Beard RW, Johnston DG. Reduced postprandial energy expenditure in women predisposed to type 2 diabetes. Diabet Med. 1994 Jul;11(6):545-50. doi: 10.1111/j.1464-5491.1994.tb02033.x. PMID 7955970
- [Background] Robinson S, Chan SP, Spacey S, Anyaoku V, Johnston DG, Franks S. Postprandial thermogenesis is reduced in polycystic ovary syndrome and is associated with increased insulin resistance. Clin Endocrinol (Oxf). 1992 Jun;36(6):537-43. doi: 10.1111/j.1365-2265.1992.tb02262.x. PMID 1424179
- [Background] Segal KR, Pi-Sunyer FX. Exercise, resting metabolic rate, and thermogenesis. Diabetes Metab Rev. 1986;2(1-2):19-34. doi: 10.1002/dmr.5610020102. No abstract available. PMID 3522143
- [Background] Forbes S, Robinson S, Parker KH, Macdonald IA, McCarthy MI, Johnston DG. The thermic response to food is related to sensitivity to adrenaline in a group at risk for the development of type II diabetes. Eur J Clin Nutr. 2009 Nov;63(11):1360-7. doi: 10.1038/ejcn.2009.91. Epub 2009 Aug 26. PMID 19707224
- [Background] Simonsen L, Bulow J, Astrup A, Madsen J, Christensen NJ. Diet-induced changes in subcutaneous adipose tissue blood flow in man: effect of beta-adrenoceptor inhibition. Acta Physiol Scand. 1990 Jun;139(2):341-6. doi: 10.1111/j.1748-1716.1990.tb08932.x. PMID 1973329
- [Background] Astrup A, Simonsen L, Christensen NJ. Effects of beta-adrenergic blockade on meal-induced thermogenesis. Clin Physiol. 1990 May;10(3):305-7. doi: 10.1111/j.1475-097x.1990.tb00100.x. No abstract available. PMID 1972046
- [Background] Ikeda K, Fujimoto S, Goto M, Yamada C, Hamasaki A, Shide K, Kawamura T, Inagaki N. Impact of endogenous and exogenous insulin on basal energy expenditure in patients with type 2 diabetes under standard treatment. Am J Clin Nutr. 2011 Dec;94(6):1513-8. doi: 10.3945/ajcn.111.017889. Epub 2011 Nov 2. PMID 22049163
- [Background] Griffith RC, Scharp DW, Hartman BK, Ballinger WF, Lacy PE. A morphologic study of intrahepatic portal-vein islet isografts. Diabetes. 1977 Mar;26(3):201-14. doi: 10.2337/diab.26.3.201. PMID 402300
- [Background] Andersson A, Korsgren O, Jansson L. Intraportally transplanted pancreatic islets revascularized from hepatic arterial system. Diabetes. 1989 Jan;38 Suppl 1:192-5. doi: 10.2337/diab.38.1.s192. PMID 2492004
- [Background] Meier JJ, Hong-McAtee I, Galasso R, Veldhuis JD, Moran A, Hering BJ, Butler PC. Intrahepatic transplanted islets in humans secrete insulin in a coordinate pulsatile manner directly into the liver. Diabetes. 2006 Aug;55(8):2324-32. doi: 10.2337/db06-0069. PMID 16873697
- [Background] Barton FB, Rickels MR, Alejandro R, Hering BJ, Wease S, Naziruddin B, Oberholzer J, Odorico JS, Garfinkel MR, Levy M, Pattou F, Berney T, Secchi A, Messinger S, Senior PA, Maffi P, Posselt A, Stock PG, Kaufman DB, Luo X, Kandeel F, Cagliero E, Turgeon NA, Witkowski P, Naji A, O'Connell PJ, Greenbaum C, Kudva YC, Brayman KL, Aull MJ, Larsen C, Kay TW, Fernandez LA, Vantyghem MC, Bellin M, Shapiro AM. Improvement in outcomes of clinical islet transplantation: 1999-2010. Diabetes Care. 2012 Jul;35(7):1436-45. doi: 10.2337/dc12-0063. PMID 22723582
- [Background] Shapiro AM. Islet transplantation in type 1 diabetes: ongoing challenges, refined procedures, and long-term outcome. Rev Diabet Stud. 2012 Winter;9(4):385-406. doi: 10.1900/RDS.2012.9.385. Epub 2012 Dec 28. PMID 23804275
- [Background] Gabe SM, Bjarnason I, Tolou-Ghamari Z, Tredger JM, Johnson PG, Barclay GR, Williams R, Silk DB. The effect of tacrolimus (FK506) on intestinal barrier function and cellular energy production in humans. Gastroenterology. 1998 Jul;115(1):67-74. doi: 10.1016/s0016-5085(98)70366-x. PMID 9649460
- [Background] Ersoy A, Baran B, Ersoy C, Kahvecioglu S, Akdag I. Calcineurin inhibitors and post-transplant weight gain. Nephrology (Carlton). 2008 Oct;13(5):433-9. doi: 10.1111/j.1440-1797.2008.00916.x. Epub 2008 Mar 5. PMID 18331443
- [Background] Yi CX, la Fleur SE, Fliers E, Kalsbeek A. The role of the autonomic nervous liver innervation in the control of energy metabolism. Biochim Biophys Acta. 2010 Apr;1802(4):416-31. doi: 10.1016/j.bbadis.2010.01.006. Epub 2010 Jan 11. PMID 20060897
- [Background] Chang HR, Lin CC, Lian JD. Early experience with enteric-coated mycophenolate sodium in de novo kidney transplant recipients. Transplant Proc. 2005 Jun;37(5):2066-8. doi: 10.1016/j.transproceed.2005.03.105. PMID 15964340
- [Background] Geddes J, Wright RJ, Zammitt NN, Deary IJ, Frier BM. An evaluation of methods of assessing impaired awareness of hypoglycemia in type 1 diabetes. Diabetes Care. 2007 Jul;30(7):1868-70. doi: 10.2337/dc06-2556. Epub 2007 Apr 6. No abstract available. PMID 17416785
- [Background] Armuzzi A, Candelli M, Zocco MA, Andreoli A, De Lorenzo A, Nista EC, Miele L, Cremonini F, Cazzato IA, Grieco A, Gasbarrini G, Gasbarrini A. Review article: breath testing for human liver function assessment. Aliment Pharmacol Ther. 2002 Dec;16(12):1977-96. doi: 10.1046/j.1365-2036.2002.01374.x. PMID 12452932
- [Background] Cox DJ, Irvine A, Gonder-Frederick L, Nowacek G, Butterfield J. Fear of hypoglycemia: quantification, validation, and utilization. Diabetes Care. 1987 Sep-Oct;10(5):617-21. doi: 10.2337/diacare.10.5.617. PMID 3677982
- [Background] DeVries JH, Snoek FJ, Kostense PJ, Masurel N, Heine RJ; Dutch Insulin Pump Study Group. A randomized trial of continuous subcutaneous insulin infusion and intensive injection therapy in type 1 diabetes for patients with long-standing poor glycemic control. Diabetes Care. 2002 Nov;25(11):2074-80. doi: 10.2337/diacare.25.11.2074. PMID 12401759
- [Background] Aleman-Mateo H, Huerta RH, Esparza-Romero J, Mendez RO, Urquidez R, Valencia ME. Body composition by the four-compartment model: validity of the BOD POD for assessing body fat in Mexican elderly. Eur J Clin Nutr. 2007 Jul;61(7):830-6. doi: 10.1038/sj.ejcn.1602597. Epub 2007 Jan 17. PMID 17228350
- [Background] Hansen AL, Carstensen B, Helge JW, Johansen NB, Gram B, Christiansen JS, Brage S, Lauritzen T, Jorgensen ME, Aadahl M, Witte DR; ADDITION-Denmark Steering Committee. Combined heart rate- and accelerometer-assessed physical activity energy expenditure and associations with glucose homeostasis markers in a population at high risk of developing diabetes: the ADDITION-PRO study. Diabetes Care. 2013 Oct;36(10):3062-9. doi: 10.2337/dc12-2671. Epub 2013 Jun 11. PMID 23757430
- [Background] Melanson EL Jr, Freedson PS. Physical activity assessment: a review of methods. Crit Rev Food Sci Nutr. 1996 May;36(5):385-96. doi: 10.1080/10408399609527732. PMID 8725670
- [Background] Wilson HJ, Dickinson F, Hoffman DJ, Griffiths PL, Bogin B, Varela-Silva MI. Fat free mass explains the relationship between stunting and energy expenditure in urban Mexican Maya children. Ann Hum Biol. 2012 Sep;39(5):432-9. doi: 10.3109/03014460.2012.714403. Epub 2012 Oct 4. PMID 23035655
- [Background] Lutomski JE, van den Broeck J, Harrington J, Shiely F, Perry IJ. Sociodemographic, lifestyle, mental health and dietary factors associated with direction of misreporting of energy intake. Public Health Nutr. 2011 Mar;14(3):532-41. doi: 10.1017/S1368980010001801. Epub 2010 Aug 16. PMID 20707944
- [Background] Jia X, Craig LC, Aucott LS, Milne AC, McNeill G. Repeatability and validity of a food frequency questionnaire in free-living older people in relation to cognitive function. J Nutr Health Aging. 2008 Dec;12(10):735-41. doi: 10.1007/BF03028622. PMID 19043649
- [Background] Jequier E, Felber JP. Indirect calorimetry. Baillieres Clin Endocrinol Metab. 1987 Nov;1(4):911-35. doi: 10.1016/s0950-351x(87)80011-3. PMID 3330435
- [Background] Kousta E, Parker KH, Lawrence NJ, Penny A, Millauer BA, Anyaoku V, Mulnier H, Forster DC, MacDonald IA, Robinson S, McCarthy MI, Johnston DG. Delayed metabolic and thermogenic response to a mixed meal in normoglycemic European women with previous gestational diabetes. J Clin Endocrinol Metab. 2002 Jul;87(7):3407-12. doi: 10.1210/jcem.87.7.8698. PMID 12107258
- [Background] Speakman J. Doubly-labelled water: theory and practice. . New York N, editor: Kluwer Academic Publishers; 1997.
- [Background] Stewart, A., Marfell-Jones, M., Olds, T., & Ridder, J.H. (2011). International standards for anthropometric assessment. Lower Hutt, New Zealand: International Society for the Advancement of Kinanthropometry